CLINICAL TRIAL: NCT06337747
Title: A Prospective, Randomized-controlled Trial Comparing Superficial Injections With Poly-L-Lactic Acid in the Temporal Fossa Versus Extended Temporal Fossa + Hairline
Brief Title: Comparing Injections With Poly-L-Lactic Acid in the Temporal Fossa vs. Extended Temporal Fossa + Hairline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-2023-PLLA
Record Dates: First submitted 2023-05-23; First posted 2024-03-29 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2023-06

CONDITIONS: Aging
Keywords: Temple; Poly-L-lactic acid; Aesthetic; Dermal fillers

STUDY DESIGN:
Intervention Model Description: A prospective, randomized-controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional technique (Active Comparator)
  Interventions: Device: Traditional technique
- Extended technique (Experimental)
  Interventions: Device: Experimental technique

INTERVENTIONS:
Device: Traditional technique — Subjects randomized to the traditional technique will receive 3cc of PLLA (per side, per treatment) in the anterior temporal region.
  Arms: Traditional technique
Device: Experimental technique — Subjects randomized to the extended technique will receive 3cc of PLLA (per side, per treatment) in the anterior temporal region, as well as 2cc (per side, per treatment) in the posterior (i.e., behind the hairline) temporal region.
  Arms: Extended technique

SUMMARY:
The use of poly-L-Lactic acid (PLLA) has demonstrated significant improvement in multiple facial and body regions. Its use in the temporal fossa is the ideal location to demonstrate its impact on neocollagenesis given its distinct anatomic boundaries. Furthermore, the fact that the lateral boundary of the temporal region can extend into the hairline allows for a graded effect to be measured. Therefore, this study aims to extend these findings by evaluating the efficacy and safety of two injection techniques for volumizing temporal hollows.

DETAILED DESCRIPTION:
Non-invasive treatment of volume loss is one of the most common aesthetic treatments performed worldwide. Poly-L-lactic acid has been used as a skin filler since 1999 in Europe and since 2004 in the United States (Vlegger, 2014), as well as in several medical areas for over three decades (Chen, 2014; Vlegger, 2006) In addition, poly-L-lactic acid is widely used in several countries for facial rejuvenation, with extensive documentation of their efficacy and safety in this context (Vlegger, 2014). Sculptra® Aesthetic is an injectable implant containing microparticles of poly-L-lactic acid, carboxymethylcellulose, non-pyrogenic mannitol and sterile water for injection. Sculptra® Aesthetic is available in 367.5 mg dose vials and is to be reconstituted prior to use by the addition of 8 mL of sterile water + 1mL xylocaine for injection to form a sterile nonpyrogenic suspension.

Sculptra® Aesthetic is indicated for increasing the volume of depressed areas, particularly to correct skin depressions such as in skin creases, wrinkles, folds, scars and for skin aging. It is also suitable for large volume corrections of the signs of facial fat loss (lipoatrophy). Poly-L-lactic acid is capable of increasing the dermal tissue through stimulating production of collagen, contributing to filling, volumizing in the treated area (Lowe, 2006; Vlegger, 2014). Unlike other skin fillers that promote volume increase shortly after injection (e.g., HA), poly-L-lactic acid exerts its effect over the course of a few weeks. This effect is usually visible after two months and noticeable up to two years after treatment (Chen, 2014; Vlegger, 2006; Vlegger, 2014)

The use of poly-l-lactic acid (PLLA) has demonstrated significant improvement in multiple facial and body regions. Its use in the temporal fossa is the ideal location to demonstrate its impact on neocollagenesis given its distinct anatomic boundaries. Furthermore, the fact that the lateral boundary of the temporal region can extend into the hairline allows for a graded effect to be measured. Therefore, this study aims to extend these findings by evaluating the efficacy and safety of two injection techniques for volumizing temporal hollows.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must voluntarily sign and date an informed consent, approved by an independent ethics committee, prior to the initiation of any screening or study-specific procedures.
* Subjects must be adult male or female, at least 18 years old.
* Subjects must be willing and able to comply with procedures required in the protocol.
* Subjects must be in good health as per investigator's judgment based on medical history.
* Subjects must have mild to severe temporal fossa hollowing.
* Subjects must not have uncontrolled systemic disease.
* Subjects do not present with or have a history of any medical condition that may place the subject at increased risk following exposure to PLLA or interfere with the study evaluation, including:

  * History of facial nerve palsy.
  * Infection or dermatological condition at the treatment injection sites.
  * Marked facial asymmetry, dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, or excessively photodamaged skin.
  * Any eyebrow or eyelid ptosis at Baseline as determined by the investigator.
* Subjects do not have history of clinically significant medical conditions or any other reason that the investigator determines would interfere with the subject's participation in this study or would make the subject an unsuitable candidate to receive study drug.
* Subjects do not have history of an allergic reaction or significant sensitivity to constituents of the study drug (or its excipients).
* Subjects must not have tattoos, jewelry, or clothing which obscure the temporal region and cannot be removed.
* Subjects do not have anticipated need for surgery or overnight hospitalization during the study.
* Subjects do not have a history of surgical procedures on forehead and/or periorbital areas or affecting these areas including any lifting procedure (e.g., facial lift, suture lift, thread lift, brow lift, eyelid and/or eyebrow surgery).
* Subjects do not have history of periorbital or upper-facial treatment with semi- permanent or permanent soft tissue fillers (e.g., poly-L-lactic acid, polyalkylimide, polymethylmethacrylate, polytetrafluoroethylene, and silicone), synthetic implantation and/or autologous fat transplantation.
* One month prior to enrolment: Subjects do not have any periorbital or upper-facial cosmetic procedures with superficial-to-medium resurfacing/planning (e.g., microdermabrasion, dermaplaning, dermabrasion), chemical peels (e.g., glycolic acid, trichloroacetic acid and phenol), or nonablative energy-based facial treatments (e.g., radiofrequency, ultrasound, electromagnetic, laser, light).
* Three months prior to enrolment: Subjects do not have ablative energy-based facial treatments or permanent make-up.
* Twelve months prior to enrolment: any periorbital or upper-facial treatment with nonpermanent soft tissue fillers (e.g., hyaluronic acid-based fillers, calcium hydroxylapatite, and collagen-based fillers).
* Subjects with known active COVID infection within 14 days of treatment.
* Female subjects of child-bearing potential must have a negative urine pregnancy test prior to any dose of study product.
* Female subjects of childbearing potential must practice at least 1 protocol-specified method of birth control that is effective from Baseline through at least 30 days after the last dose or until the end of study, whichever is longer. Female subjects of non-childbearing potential do not need to use birth control.
* Female subjects that are not pregnant or breastfeeding and are not considering becoming pregnant or donating eggs during the study or for approximately 30 days after the last dose of study drug or until the end of study, whichever is longer.
* Subjects must not have been treated with any investigational drug within 30 days prior to the first dose of study drug or is currently enrolled in another clinical study.
* Using or planning to initiate restrictive diets that could result in extreme fluctuations in weight (i.e., +/- 10 lbs), at investigator's discretion.
* Using or planning to initiate the use of supplements for weight loss.
* Using or have used within the previous 3 months drugs such as corticosteroids, immunosuppressants, anticoagulants or other collagen-production inhibitors.
* Initiated use of hormones or change in dose of hormonal replacement therapy within 3 months, due to possible implications on weight.
* Sculptra® Aesthetic should not be used in patients with known history of or susceptibility to keloid formation or hypertrophic scarring.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
To access the efficacy of the tradition and experimental technique | Baseline to Week 7, Week 14, Week 20, Week 28, Week 38
  To assess the efficacy of poly-l-lactic acid for volumization of the temporal fossae, between standard and extended techniques at all follow-up visits.

SECONDARY OUTCOMES:
To access the safety of the tradition and experimental technique | Baseline to Week 7, Week 14, Week 20, Week 28, Week 38
  To assess the safety of poly-l-lactic acid for volumization of the temporal fossae between the standard and extended techniques, at all visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Erevna Innovations Inc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen HH, Javadi P, Daines SM, Williams EF 3rd. Quantitative assessment of the longevity of poly-L-lactic acid as a volumizing filler using 3-dimensional photography. JAMA Facial Plast Surg. 2015 Jan-Feb;17(1):39-43. doi: 10.1001/jamafacial.2014.867. PMID 25340593
- [Background] Lowe NJ. Dispelling the myth: appropriate use of poly-L-lactic acid and clinical considerations. J Eur Acad Dermatol Venereol. 2006 May;20 Suppl 1:2-6. doi: 10.1111/j.1468-3083.2006.01515.x. PMID 16643417
- [Background] Vleggaar D. Soft-tissue augmentation and the role of poly-L-lactic acid. Plast Reconstr Surg. 2006 Sep;118(3 Suppl):46S-54S. doi: 10.1097/01.prs.0000234846.00139.74. PMID 16936544
- [Background] Vleggaar D, Fitzgerald R, Lorenc ZP. Composition and mechanism of action of poly-L-lactic acid in soft tissue augmentation. J Drugs Dermatol. 2014 Apr;13(4 Suppl):s29-31. PMID 24719074
- [Background] Ali A. Contouring of the gluteal region in women: enhancement and augmentation. Ann Plast Surg. 2011 Sep;67(3):209-14. doi: 10.1097/SAP.0b013e318206595b. PMID 21587056